CLINICAL TRIAL: NCT06659211
Title: Effectiveness of Mentalization-based Therapy (MBT) as Part of a Stepped Mental Health Care in Finland - a Pilot Study
Brief Title: Effectiveness of Mentalization-based Therapy (MBT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240/2024
Record Dates: First submitted 2024-10-02; First posted 2024-10-26 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-10

CONDITIONS: Severe Mental Illness
Keywords: mentalization, MBT, severe mental disorder, therapy, psychotherapeutic
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mentalisation-Based Therapy (Experimental): MBT is conducted according to the treatment manual developed by Bateman & Fonagy. Patients are offered weekly individual sessions with an MBT therapist for 12 months.
  Interventions: Behavioral: Mentalisation-Based Therapy
- Treatment as usual (Active Comparator): The TAU group will receive treatment as usual, which in mental health services might include medication, supportive counseling, short therapy, and other limited psychotherapeutic treatments such as DKT. There is no requirement for a frequency of visits for the usual psychiatric care of the TAU group, as this would not be realistic in the current service system.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Mentalisation-Based Therapy — MBT is conducted according to the treatment manual developed by Bateman & Fonagy. Patients are offered weekly individual sessions with an MBT therapist for 12 months.
  Arms: Mentalisation-Based Therapy
Other: Treatment as Usual (TAU) — The TAU group will receive treatment as usual, which in mental health services might include medication, supportive counseling, short therapy, and other limited psychotherapeutic treatments such as DKT. There is no requirement for a frequency of visits for the usual psychiatric care of the TAU group, as this would not be realistic in the current service system, and the usual treatment would not be the usual treatment currently provided.
  Arms: Treatment as usual

SUMMARY:
The effects of psychological treatment, mentalization-based therapy, will be studied among persons with mental disorders seeking help from mental health care services.

DETAILED DESCRIPTION:
Background: Mentalization-based therapy (MBT) has a growing evidence base as a group treatment, and research on MBT as an individual treatment is needed. This study will provide crucial new information on its effectiveness and usability in everyday patient care.

Methods: The study design will be an non-randomized clinical pilot study. We will study the effectiveness of MBT and analyze which factors are associated with better effectiveness. The length of intervention will be 12 months. The primary outcome measure is the change in psychological symptoms and well-being from the beginning to the end of MBT treatment, measured by CORE-OM. Secondary outcomes include several measures of symptoms, functioning, quality of life, and mentalization. Outcomes will be assessed at 6, 12 and 18 months. The study group will comprise of 64 patients receiving MBT. For comparison, patient group (n=64) with similar characteristics (age, gender, diagnosis) receiving treatment as usual (TAU) in psychiatric services will be ascertained from medical records, and their outcomes after 12 months of treatment will be compared to that of MBT -group.

Intervention / Treatment: Behavioral: Mentalization-based treatment/therapy

Participation criteria: Patients are not strictly limited to a specific disease/diagnostic group. This choice has been made because there is an increasing need in the mental health care for the treatment and therapy of this multi-symptom and severely symptomatic patient group, which also makes the results of the study more applicable to a real life. Patients will be selected for the MBT and TAU based on inclusion and exclusion criteria and patients preference. In addition, the selection to MBT will be made by a trained MBT therapist, who will assess the patient's suitability for MBT (e.g., patient willing to engage in active psychotherapeutic work, interested in the inner world of experience, willing to work interactively).

ELIGIBILITY:
Inclusion Criteria:

MBT Group:

* Age 18-64 years.
* Severe psychological symptoms, decreased functioning ability for long-term
* Challenges with interpersonal relationships and emotional regulation
* Patients willing to receive MBT
* At least two of the following:

  * Depression (diagnosis codes: F31.3-F31.5, F32.0-F32.9, F33.3-F33.9, F34.1) or anxiety disorder (diagnosis codes: F40-F48)
  * Trauma background either as diagnosis or as need for treatment
  * Signs of personality disorder (suspected or diagnosed)

TAU group:

* Age 18-64 years.
* Severe psychological symptoms, decreased functioning ability for long-term
* Challenges with interpersonal relationships and emotional regulation
* At least two of the following

  * Depression (diagnosis codes: F31.3-F31.5, F32.0-F32.9, F33.3-F33.9, F34.1) or anxiety disorder (diagnosis codes: F40-F48)
  * Trauma background either as diagnosis or as need for treatment
  * Signs of personality disorder (suspected or diagnosed)

Exclusion Criteria:

MBT Group:

* Active substance use disorder (i.e., intoxication F1x.0, active dependence F1x.24, Continuous use F1x.25), a physiological withdrawal state F1x.3 and F1x.4, or psychotic disorder F1x.5).
* Acute psychosis (defined as the recent onset of severe psychotic symptoms that interfere with functioning and are not yet in a therapeutic state. Non-acute psychotic symptoms are not exclusionary)
* Disorder requiring inpatient treatment
* Previously received MBT
* Currently receiving psychotherapeutic treatment (previous psychotherapeutic treatment is not an exclusion)

The exclusion criteria, therefore, do not exclude psychotic disorders or any other psychiatric illness (except substance abuse disorders).

TAU group:

* Active substance use disorder (i.e., intoxication F1x.0, active dependence F1x.24, Continuous use F1x.25), a physiological withdrawal state F1x.3 and F1x.4, or psychotic disorder F1x.5).
* Acute psychosis (defined as the recent onset of severe psychotic symptoms that interfere with functioning and are not yet in a therapeutic state. Non-acute psychotic symptoms are not exclusionary)
* Disorder requiring inpatient treatment
* Previously received MBT
* Intensive psychotherapy (e.g. rehabilitative psychotherapy or similar weekly long-term psychotherapy)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM) | baseline, 6, 12 and 18 months
  A self-report measure of psychological distress and symptoms. Higher scores indicates worse outcomes. Includes four main domains: wellbeing, problems, functioning and risk (to self or others).
  Based on detailed instructions on calculating the scores, clinical score minimun 0 and maximum 40.

SECONDARY OUTCOMES:
The Big Five Inventory-2 Extra-Short Form (BFI-2-XS) | baseline, 6, 12 and 18 months
  questionnaire assessing personality
the Inventory of Interpersonal Problems (IIP-32) | baseline, 6, 12 and 18 months
  Questionnaire on interpersonal problems
Experiences in Close Relationships Short version (ECR-S) | baseline, 6, 12, and 18 months
  Measures experiences in close relationships
Rosenberg Self-Esteem Scale (RSE) | baseline, 6, 12, and 18 months
  Questionnaire on self-esteem
Emotion Regulation Questionnaire (ERQ) | baseline, 6, 12 and 18 months
  Measure of emotion regulation
The Certainty About Mental States Questionnaire (CAMSQ) | baseline, 6, 12 and 18 months
  Questionnaire on perceived capacity of mentalising oneself and others.
The Reflective Functioning Questionnaire (RFQ) | baseline, 6, 12 and 18 months
  a brief measure of reflective functioning, i.e. mentalizing
Quality of life | baseline, 6, 12 and 18 months
  WHO 1 question
The Montgomery-Åsberg Depression Rating Scale (MADRS) | baseline, 12 months
  Interview based rating of depression symptoms and their severity. Minimum: 0 Maximum: 60 Higher scores indicate more severe symptoms.
Social and Occupational Functioning Assessment Scale (SOFAS) | baseline, 12 months
  Clinician/investigator rated measure of social and occupational functioning. Minimum value: 0 (Inadequate information), 1 (worst functioning, unable to function, persistent inability) Maximum value: 100 (Superior functioning in a wide range of activities)
Clinical Global Impression- Severity scale (CGI-S) | baseline, 12 months
  Clinical Global Impression of the severity of illness. Minimum value: 1 (normal, not at all ill) Maximum value: 7 (amongst the most severely ill)
Working Alliance Inventory (WAI) | baseline, 6 and 12 months
  Questionnaire on therapeutic alliance. Higher scores indicate better alliance.
Suicidality | from baseline to 18 months
  from questionnaires and medical records
Patient experiences of the treatment | 6 and 12 months
  questions on how the patient has experienced the intervention, and if he/she has experienced the treatment as beneficial
Experiences of recovery | 12 and 18 months
  Questions on experience of change of health status and recovery

OTHER OUTCOMES:
Physical symptoms and illnesses | from baseline to 12 months
  Information collected from the medical records. Data on physical symptoms or diagnosed physical illnesses, that the patient complains or seeks help will be collected from the medical records (visits to mental health care and somatic care).
Need of psychiatric services | from baseline to 12 months
  Number of outpatient, inpatient and emergency visits. Data from medical records.
Use of medication | from baseline to 12 months
  Use of psychiatric medications. Data from medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No